CLINICAL TRIAL: NCT01778894
Title: Mathematical Modeling to Determine Basic Muscle Properties in the Failing Heart
Status: Terminated | Type: Observational
Why Stopped: Administratively closed because no Continuing Review submitted
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0623-12-EP
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Diastolic Heart Failure
Keywords: Diastolic Dysfunction, Diastolic Heart Failure, Diastolic; Echocardiography
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Murmurs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Healthy controls with no history of heart disease or heart failure. Subjects will undergo a medical history review and 1 echocardiograph procedure.
- >Grade 2 Diastolic Dysfunction: Diastolic Heart Failure, > Grade II (NYHA functional class) and/or > Grade II Diastolic Dysfunction as evaluated by echocardiography

SUMMARY:
According to the most recent information released by the American Heart Association, heart failure affects 5.8 million Americans and over 23 million people worldwide. In particular, diastolic heart failure (DHF) has emerged in approximately half of those suffering from heart disease and has become a major public health problem for many reasons, including the complexity of the disease, lack of effective drugs/therapies, requirement of invasive tests to diagnose and monitor DHF, and the absence of a suitable scientific model to study the disease. Scientists and physicians alike still do not fully understand what happens to the muscles in the heart (myocardium) patients who present with diastolic dysfunction or DHF. Therefore, the medical field is in need of an accurate model that can evaluate how diastolic dysfunction leads to heart failure and what happens at a cellular level as this disease emerges and progresses.

DETAILED DESCRIPTION:
Our group has developed a mathematical model of the heart that gathers data from a procedure called an echocardiograph (echo) to analyze how muscles in the heart are functioning. This model incorporates how the heart muscle functions on a cellular level along with the overall functionality of the heart.

We hypothesize that this model will measure the specific properties of the heart muscle that affect their ability to contract and relax. This study will determine whether these properties will be different in patients with DHF compared to healthy controls. We also propose that these abnormalities in the heart muscle will correlate with the patient's degree of heart failure and their prognosis when doctors evaluate using standard clinical tests.

This study will be conducted at the University of Nebraska Medical Center (UNMC). 40 subjects will be enrolled, 20 healthy controls with no history of heart disease and 20 subjects who have been diagnosed with diastolic heart failure. Healthy controls will be required to undergo 1 echocardiograph procedure at UNMC. Subjects diagnosed with DHF will be required to undergo 6 echocardiograph procedure over the course of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 19 years of age or older
* Control subjects must have no prior history or current signs of heart disease.
* Subjects with heart failure must meet one or more of the following criteria:
* Documented Diastolic Heart Failure, Grade II or greater (via NYHA functional class)
* Grade II or greater Diastolic Dysfunction by echocardiographic evaluation

Exclusion Criteria:

* Subjects under the age of 19 or unable to give consent will be excluded from this study.
* Greater than mild valvular disease
* Prior valve repair/replacement

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal controls will be recruited from the Omaha community. Subjects with Diastolic Heart Dysfunction and/or Failure will be selected from The University of Nebraska Medical Center Heart Clinic or from The Nebraska Medical Center Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
The longitudinal assessment of myocardial properties in subjects with Diastolic Heart Failure. | 2 years
  Our mathematical model of the heart integrates the cellular mechanisms of sarcomere dynamics with the overall functional properties of the ventricle. Utilizing specific measurements captured by echo, estimates of basic muscle properties in subjects suffering from DHF will be compared to observed properties. Echo measurements will be taken at baseline and 2 weeks, 4 months, 8 months, 1 year, and 2 years following therapy.

SECONDARY OUTCOMES:
Correlation of observed muscle properties to clinical outcomes/status. | 2 years
  Clinical outcome measurements, including hospitalizations, New York Heart Association (NYHA) class, and mortality, will be collected to determine effectiveness of current therapy for diastolic heart failure. By tracking patient outcomes and measured clinical endpoints, the degree of material parameter abnormality affecting clinical outcomes of subjects will be tested using multivariate regression with the material parameters derived from the model. The dependent variables and covariates such as age, sex, ejection fraction, presence of co-morbidities such as coronary artery disease, diabetes, and hypertension will also be included in the analysis.
Validation of the developing mathematical model using the data points collected from echocardiographic procedures | 1 baseline echocardiograph
  An optimization driver program that controls the parameter estimation has been developed and will be validated. To estimate unknown material parameters, multiple forward model simulations are obtained to estimate the partial derivatives of the least squares objective function with respect to the material parameters. Best-fit parameters will be determined for each DHF patient and each control using cylindrical, spherical and ellipsoidal models. Each of these parameters represents a unique aspect of sarcomere and ventricular matrix constitutive behavior. Best-fit material parameters for each patient will be compared with those obtained from the control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Moulton J Moulton, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kass DA, Bronzwaer JG, Paulus WJ. What mechanisms underlie diastolic dysfunction in heart failure? Circ Res. 2004 Jun 25;94(12):1533-42. doi: 10.1161/01.RES.0000129254.25507.d6. PMID 15217918
- [Background] Paulus WJ, Tschope C, Sanderson JE, Rusconi C, Flachskampf FA, Rademakers FE, Marino P, Smiseth OA, De Keulenaer G, Leite-Moreira AF, Borbely A, Edes I, Handoko ML, Heymans S, Pezzali N, Pieske B, Dickstein K, Fraser AG, Brutsaert DL. How to diagnose diastolic heart failure: a consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology. Eur Heart J. 2007 Oct;28(20):2539-50. doi: 10.1093/eurheartj/ehm037. Epub 2007 Apr 11. PMID 17428822
- [Background] Moulton MJ, Creswell LL, Actis RL, Myers KW, Vannier MW, Szabo BA, Pasque MK. An inverse approach to determining myocardial material properties. J Biomech. 1995 Aug;28(8):935-48. doi: 10.1016/0021-9290(94)00144-s. PMID 7673261